CLINICAL TRIAL: NCT00002753
Title: PROTOCOL FOR A PHASE I STUDY OF INTRACYSTIC ANTI-TENASCIN MONOCLONAL ANTIBODY 131I 81C6 IN THE TREATMENT OF PATIENTS WITH RECURRENT CYSTIC GLIOMAS
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Recurrent Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000064689; DUMC-1965-98-12R7; DUMC-1752-96-12R5; DUMC-1775-95-12R4; DUMC-1860-97-12R6; NCI-H96-0008
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood supratentorial ependymoma; recurrent childhood brain tumor; recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult myxopapillary ependymoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult ependymoblastoma; recurrent childhood cerebral astrocytoma; recurrent childhood ependymoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Ependymoma; Oligodendroglioma; Glioma; Neuroectodermal Tumors, Primitive; Familial ependymoma; Gliosarcoma

INTERVENTIONS:
Radiation: iodine I 131 monoclonal antibody 81C6

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to determine the effectiveness of monoclonal antibody in treating patients with recurrent gliomas.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxic effects of intracystic administration of iodine-131-labeled anti-tenascin monoclonal antibody 81C6. II. Identify any objective therapeutic responses to this treatment in patients with recurrent cystic anaplastic gliomas.

OUTLINE: Radioimmunotherapy. Iodine-131-Labeled Anti-Tenascin Monoclonal Antibody 81C6, 131I-81C6.

PROJECTED ACCRUAL: Three to six patients will be entered at each dose studied.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed supratentorial anaplastic glioma with a recurrent cyst requiring aspiration for symptom control Measurable cystic lesion confirmed by contrast-enhanced CT or MRI At least 3 months since radiotherapy to site of measurable disease unless unequivocal evidence of tumor progression Neoplastic cell reactivity with tenascin demonstrated by immunohistology with either a polyclonal rabbit antibody or a monoclonal murine antibody

PATIENT CHARACTERISTICS: Age: 3 and over Performance status: Karnofsky 50-100% Hematopoietic: Absolute neutrophil count greater than 1,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL AST less than 1.5 times normal Alkaline phosphatase less than 1.5 times normal Renal: Creatinine less than 1.2 mg/dL Other: Negative pregnancy test Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 6 weeks since antineoplastic chemotherapy unless unequivocal evidence of tumor progression Endocrine therapy: Corticosteroids allowed if at lowest possible dose and dose stable for at least 10 days prior to entry Radiotherapy: See Disease Characteristics Surgery: Not specified

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 1991-11; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darell D. Bigner, MD, PhD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States